CLINICAL TRIAL: NCT00192543
Title: A Clinical Trial of Fish and Fruit to Improve Survival of Aboriginal People With End Stage Renal Disease
Brief Title: The Fish and Fruit Study: Trial of Fish and Fruit to Improve Survival of Aboriginal People With End Stage Renal Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: The George Institute (Other); Northern Territory Government of Australia (Other Government)
Responsible Party: Gurmeet Singh, Menzies School of Health Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 283304
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2009-03

CONDITIONS: Cardiovascular Diseases
Keywords: dialysis; omega-3 fatty acids; antioxidants; cardiovascular markers; Mortality; End-stage renal disease
MeSH Terms: conditions — Cardiovascular Diseases; Kidney Failure, Chronic | interventions — Fruit; Diet; In Situ Hybridization, Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- case (Active Comparator): diet of fish and fruit addition compared to regular diet
  Interventions: Behavioral: diet of fish and fruit; Behavioral: diet only
- control (Placebo Comparator): regular diet
  Interventions: Behavioral: fruit and fish; Behavioral: regular diet

INTERVENTIONS:
Behavioral: diet of fish and fruit — fish and fruit in specified quantities
  Other Names: regular diet
  Arms: case
Behavioral: fruit and fish — no drugs
  Arms: control
Behavioral: diet only — Fish and fruit
  Arms: case
Behavioral: regular diet — no change in regular diet
  Arms: control

SUMMARY:
Cardiovascular disease is the main cause of death in patients on dialysis for end stage renal disease. Omega-3 fatty acids and antioxidants have been shown to be protective in the general population. A diet of fish and fruit, which will provide the fatty acids and the antioxidants is being tried in dialysis patients to assess the effect on cardiovascular disease in this high risk group.

DETAILED DESCRIPTION:
End stage renal disease (ESRD) is a devastating disease which affects Aboriginal Australians disproportionately: The average survival time for Aboriginal people in the Northern Territory is 3.6 years from the onset of kidney failure, compared to 12.3 years for non-Aboriginal people. There has been a dramatic rise in incidence of kidney failure over the past 20 years, with the prevalence doubling every 4-5 years in many NT communities and other remote parts of Australia. Mortality for patients with ESRD is approximately 5 to 10 fold that of the general population, with heart disease accounting for approximately half of deaths.

The aims of this study are to determine whether a dietary intervention of fish and fruit three times a week will decrease cardiovascular and all-cause mortality in patients on haemodialysis in Darwin and Alice Springs . There is a strong scientific rationale for this simple dietary intervention. Fish are a rich source of omega-3 fatty acids, believed to reduce the risk of heart attack. Fruit is a good source of anti oxidants and other chemicals that may amplify the beneficial effects of fish. Participants are randomized to either control and intervention groups according to their regular days of dialysis. Nutritional and cardiovascular status will be measured at commencement of the study and then at intervals of 3, 6 and 12 months.

Strategies have been incorporated into the project design to ensure understanding, informed consent and participation of Aboriginal people in a number of domains: the participant, their family, urban and remote communities, and service providers. If successful this intervention will result in changes to the clinical management of renal patients worldwide.

ELIGIBILITY:
Inclusion Criteria:

* All patients on hemodialysis

Exclusion Criteria:

* Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2004-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Deaths due to cardiovascular disease | records continue to be checked till 2009

SECONDARY OUTCOMES:
Non-invasive cardiovascular markers: carotid intimal medial thickness | completed 2008

CONTACTS AND LOCATIONS:
Overall Officials: Kerin O'Dea, PhD, Principal Investigator — Menzies School of Health Research
Locations (1):
- Department of Health and Community Services, Darwin, Northern Territory, Australia